CLINICAL TRIAL: NCT01870089
Title: Clinical Evaluation of an Automated Knowledge-based Computer Driven System (SmartCare/PS-NIV) Designed to Automatically Adapt Pressure Support Level and Expiratory Cycling During Non Invasive Ventilation, a Feasability Study.
Brief Title: SmartCare Driven Pressure Support-Non Invasive Ventilation Feasibility Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enough data to conclude
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Prof. Philippe Jolliet, Principal investigator, University of Lausanne Hospitals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SmartCare/PS-NIV
Record Dates: First submitted 2013-05-23; First posted 2013-06-05 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Acute Respiratory Failure
Keywords: Non invasive ventilation; Computer-driven system; Acute respiratory failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study group (Experimental)
  Interventions: Device: SmartCare/PS-NIV Drägerwerk Lübeck Germany

INTERVENTIONS:
Device: SmartCare/PS-NIV Drägerwerk Lübeck Germany

SUMMARY:
Knowledge-based systems were initially developped to automatically adapt pressure support settings during invasive ventilation, and proved to be at least as efficient as experienced clinicians.

Non-invasive ventilation has become the standard of care for patients suffering from acute hypercapnic respiratory failure (ARF)and has reduced the need for endotracheal intubation in these patients, thus reducing their hospital mortality.

NIV success or failure is closely related to the tolerance of NIV treatment, which is tightly correlated to patient-ventilator synchrony. As severe asynchronies frequently occurs during NIV (namely in more than 40% of patients) and as the occurence of asynchronies is related to the use of high pressure support levels, to the presence of leaks and/or to non optimal expiratory trigger settings, very frequent ventilator settings adaptations should allow reducing patient-ventilator asynchronies but require the presence of an experienced clinician at the bedside during NIV treatment.

A computer-driven ventilator settings adaptation has the adavantage of permitting very frequent ventilator settings adaptation whithout requiring the presence of an experienced clinician at the bedside and could possibly improve patient-ventilator interaction.

The aim of the present study is to test the faisability of using the Smartcare NIV computer-driven system to automatically adapt ventilator settings during non invasive ventilation delivered because of acute respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* Acute respiratory failure requiring non invasive ventilation
* ICU patient equipped with an arterial line.

Exclusion Criteria:

* Contra-indications to NIV:
* impaired consciousness
* absence of patient cooperation
* severe hemodynamic instability
* vomiting
* facial lesions
* indication for immediate intubation
* Acute neurological problem
* Poor short term prognosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-05; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Feasibilty of using the Smartcare-NIV system to deliver non-invasive ventilation in case of acute respiratory failure. | 45 minute NIV-treatment
  The main aim of the study is to explore the feasibility of using the Smartcare-NIV system to deliver non-invasive ventilation (NIV) in case of acute respiratory failure. Practically, we will describe how the NIV tratment will go on when using the Smartcare system and report how the system automatically adapt the ventilator settings.

SECONDARY OUTCOMES:
Respiratory rate | 45 minutes
Minute ventilation | 45 minutes
Tidal volumes | 45 minutes
Leaks | 45 minutes
O2 saturation | 45 minutes
  Transcutaneous measurement
Alarms generated by the ventilator | 45 minutes
Manual ventilator settings modifications required | 45 minutes
Patient-ventilator asynchronies | 45 minutes
Blood gas analysis | 45 minutes
  Two blood gas analysis will be done, one at the beginning and one at the end of the 45-minyte NIV treatment.
Patient comfort | 45 minutes
  Patient comfort will be evaluated usuing a visual analogic scale graduated between 0 and 10.
Percentage of time spent in a predifined comfort zone. | 45 minutes
  The comfort zone will be defined as respiratory rate between 14 and 29 breaths/minunte and tidal volume between 5 and 10 ml/ kg IBW
Heart rate | 45 minutes
Blood pressure | 45 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Jolliet, Prof, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Adult Intensive Care and Burn unit, University Hospital of Lausanne, Lausanne, Switzerland